CLINICAL TRIAL: NCT02753855
Title: Pharmacokinetics of Telavancin in Normal and Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Principal Investigator, Keith A. Rodvold, Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TELAPK-2015
Record Dates: First submitted 2016-04-18; First posted 2016-04-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
MeSH Terms: interventions — telavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telavancin Administration (Experimental): Single dose of telavancin administered as a 1-hour intravenous infusion
  Interventions: Drug: Telavancin

INTERVENTIONS:
Drug: Telavancin — A single dose of telavancin as a 1-hour intravenous infusion
  Other Names: Vibativ

SUMMARY:
The purpose of this study is to characterize plasma and urinary concentrations of telavancin following intravenous administration of a single dose of telavancin in healthy subjects who are normal weight, overweight, and obese.

DETAILED DESCRIPTION:
This study is a Phase I, open-label, single-dose pharmacokinetic study in healthy adult male and female subjects. Eligible subjects will be assigned to one of four groups based on their body mass index and total body weight. Subjects will receive a single dose of telavancin depending on subject's group as a 1-hour intravenous infusion. Serial blood and urine samples will be collected over 12 hours to determine serum and urinary pharmacokinetics of telavancin. Subjects will return for blood and urine sample collection at 24 and 48 hours. Safety evaluations will be assessed throughout the study and will include physical examination, vital sign monitoring, clinical laboratory tests, monitoring of adverse events, and markers of kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects, 18 to 50 years
* Nonsmokers within the last 1 year
* Weight > 110 lbs

Exclusion Criteria:

* History of significant hypersensitivity reaction or intolerance to telavancin
* Aspartate or alanine aminotransferase > 1.5 times the upper limit of normal
* Estimated creatinine clearance <60 mL/minute and serum creatinine >1.5 mg/dL
* Female subjects who are pregnant or breast feeding
* History of alcohol or substance abuse or dependence within the last 1 year
* Use of prescription or nonprescription drugs (unless hormonal contraceptives) within 7 to 14 days prior to telavancin administration
* Participation in a clinical trials within last 30 days
* Donated blood (>500 mL) within the last 56 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number (%) of adverse events of any severity regardless of relationship to study drug | 48 hours
Area-under-the-plasma concentration-time curve (AUC0-infinity) | 48 hours
  To estimate the telavancin pharmacokinetic parameter area-under-the-plasma concentration-time curve (AUC0-infinity) after a single dose of telavancin in healthy adult participants
Maximum plasma concentration (Cmax) | 48 hours
  To estimate the telavancin pharmacokinetic parameter maximum plasma concentration (Cmax) after a single dose for intravenously dosed telavancin to healthy adult participants

CONTACTS AND LOCATIONS:
Overall Officials: Keith A. Rodvold, Pharm.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bunnell KL, Pai MP, Sikka M, Bleasdale SC, Wenzler E, Danziger LH, Rodvold KA. Pharmacokinetics of Telavancin at Fixed Doses in Normal-Body-Weight and Obese (Classes I, II, and III) Adult Subjects. Antimicrob Agents Chemother. 2018 Mar 27;62(4):e02475-17. doi: 10.1128/AAC.02475-17. Print 2018 Apr. PMID 29311094